CLINICAL TRIAL: NCT05766046
Title: Early Diagnosis of Lung Cancer of the Italian Pulmonary Screening Network (RISP): Comparative Analysis for the Use of Low Dose Computed Tomography and Promotion of Primary Prevention Interventions in Subjects at High Risk for Lung Cancer
Brief Title: Lung Cancer Prevention Screening Programme in Italy
Acronym: RISP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ugo Pastorino (Other)
Collaborators: Presidio Ospedaliero Santo Spirito, Pescara (Unknown); IRCCS Centro di Riferimento Oncologico di Basilicata, Potenza (Unknown); Azienda Ospedaliera Pugliese Ciaccio (Other); Istituto Nazionale Tumori IRCCS - Fondazione G. Pascale (Network); Azienda Ospedaliera dei Colli (Other); Azienda Ospedaliero-Universitaria di Parma (Other); IRCCS in Tecnologie Avanzate e Modelli Assistenziali in Oncologia di Reggio Emilia, Reggio Emilia (Unknown); Istituto Nazionale dei Tumori Regina Elena, Roma (Unknown); Ospedale Policlinico San Martino (Other); A.O. Ospedale Papa Giovanni XXIII (Other); Azienda Ospedaliero, Universitaria Ospedali Riuniti (Other); Azienda Provinciale per i Servizi Sanitari, Provincia Autonoma di Trento (Other); San Luigi Gonzaga Hospital (Other); Istituto Tumori Giovanni Paolo II, BARI (Unknown); Azienda Ospedaliera per l'Emergenza Canizzaro (Other); Azienda Ospedaliero-Universitaria Careggi (Other); Istituto Oncologico Veneto IRCCS (Other)
Responsible Party: Sponsor-Investigator, Ugo Pastorino, MD, Head of Thoracic Surgery Division, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Organization: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INT 292/20
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Lung Cancer; COPD (Chronic Obstructive Pulmonary Disease) With Acute Lower Respiratory Infection; Cardiovascular Diseases
Keywords: lung cancer; LDCT; cytisine; screening; smoking cessation; DOPC; cardiovascular diseases; primary prevention; secondary prevention; RCT; microRNA; biomarkers
MeSH Terms: conditions — Lung Neoplasms; Pulmonary Disease, Chronic Obstructive; Cardiovascular Diseases; Smoking Cessation | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard arm (Experimental): Volunteers with a negative baseline LDCT will repeat LDCT after the first screening with an annual interval (according to guidelines)
  Interventions: Diagnostic Test: early lung cancer detection; Other: blood test
- Risk-based arm (Experimental): Volunteers with a negative baseline LDCT will repeat LDCT after the first screening with an interval of two years.
  Interventions: Diagnostic Test: early lung cancer detection; Other: blood test

INTERVENTIONS:
Diagnostic Test: early lung cancer detection — standard treatment for early lung cancer detection with LDCT at one or two years interval
Other: blood test — blood analysis for microRNA and other biomarkers detection

SUMMARY:
This prospective randomized multicentered clinical study aims at implementing early diagnosis of lung cancer in high-risk heavy smokers in the Italian population. The main goal of the study is to develop a nationwide lung cancer prevention screening with high quality standard, similar to that of other screening programs i.e. breast, colon and cervix ongoing in Italy.

The Italian Pulmonary Screening Network (RISP) includes 18 centers, which will promote primary prevention by offering a smoking cessation program (i.e. counselling and anti-smoking cytisine-based therapy) and secondary prevention by screening volunteers with chest Low Dose Computed Tomography (LDCT). The primary objective of the study is to demonstrate the non-inferiority of a risk-based screening strategy (less intensive, every 2 years) compared to the standard annual screening, in terms of stage I/II lung cancer incidence.

Furthermore, the study aims to provide evidence whether blood biomarkers screening intervals can improve the efficiency of lung cancer screening by requiring less CT examinations while retaining the ability to diagnose lung cancer at curative state.

DETAILED DESCRIPTION:
Tobacco smoking is the most relevant cause of avoidable death in all high-income countries, including the European Union and Italy. Smoking increases the risk of dying from emphysema by 10 times, doubles that of having a stroke, and increases two to four times that of being affected by a heart attack. In addition, the carcinogenic substances contained in tobacco smoke are responsible for about 90% of lung cancers, but also for most cancers of the oral cavity, larynx and bladder. Therefore, the main causes of death attributable to tobacco smoke are cancers, cardiovascular and respiratory diseases. Lung cancer is a serious and far-reaching health problem with reduced survival after 5 years. Seventy per cent of lung cancers are at an advanced clinical stage and difficult to treat when the first symptoms occur, and a certain diagnosis is made. Lung cancer mainly affects people over the age of 50, with a peak incidence around 70-75 years. Over a third of deaths attributed to smoking are between 35 and 69 years of age. For long time it was not possible to have a certain diagnosis by diagnostic tests. Only at the end of the '90s, it became clear that computed tomography allows lung cancer to be detected at an early stage (stage I), before symptoms occur.

Large-scale randomized clinical trials (RCTs) have shown that early detection of lung cancer by CT can reduce lung cancer mortality between 20% and 39%, according to the duration of the intervention. In particular, LDCT screening has been shown to significantly reduce lung cancer mortality by 8-26% for men and 26-61% in women. International lung cancer screening guidelines, currently adopted in the United States, recommend repeating LDCT at annual intervals. However, annual chest LDCT screening has heavy economic impact and can induce radiation-related damage.

Recent studies have shown that the first LDCT screening exam provides information on individual risk thus allowing the personalization of the screening interval. In particular, there are indications that screening interval can be extended safely for low-risk individuals. For example, several studies show that individuals with a negative baseline exam have a substantially lower risk than those with a positive baseline exam. A randomized prospective assessment of risk-based screening intervals therefore has the potential to improve efficiency and reduce the economic-health impact of lung cancer screening. In fact, a personalized screening protocol has a less serious economic impact, both at the instrumental level and in terms of the commitment of the radiological staff.

In this context, the RISP network aims to promote a nationwide early diagnosis program with LDCT that reduces mortality from lung cancer, and at the same time, brings benefit in primary prevention of smoking-related diseases, such as chronic obstructive pulmonary diseases (COPD) and other cardiovascular diseases. RISP will start lung screening in a gradual and controlled way, through a network of reference centers with multidisciplinary clinical competence that provide adequate coverage of the territory, and meanwhile a level of quality fitting to the standards currently achieved in the screening of other cancers (breast, cervix, colon). A systematic screening program will also increase the percentage of lung cancer patients eligible for early-stage surgical resection from the current 25% (without screening) to 50-60%.

At baseline- each volunteer will undergo:

* a baseline questionnaire (e.g. socio-demographic, smoking habits, etc) with anti-smoking counseling program that includes cytisine-based anti-smoking therapy.
* blood sampling for the assessment of the inflammatory and metabolic profile (i.e. bio-markers) (optional)
* evaluation of respiratory function and measurement of carbon monoxide (CO)
* chest LDCT without contrast
* anthropometric evaluation (e.g. weight, height, BMI, etc)

Follow-up- each randomized volunteer will undergo:

* clinical examinations of LDCT
* blood sampling and CO after 12 months of follow-up or 24 months depending on the arm to which they belong.

Imaging will be performed by volumetric acquisition with a computed tomography scanner equipped with advanced technology hardware and software, including an AI-based second reading that will be validated by a radiologists panel.

All data will be entered into a password-protected database. The protection of the identity of the subjects will be guaranteed by assigning unique participation numbers specific to the study. In a separate database, accessible only by the principal investigator or assigned team members, the unique identification number can be linked to participants' names and addresses for the purposes of local and central administrative processes such as scheduling scans, sending invitation letters, sending screening results and questionnaires for topics, and collecting follow-up information. All volunteer samples and paper/electronic files will be destroyed 15 years after completion of the study.

Participants are assured that no personal data will be published in articles, reports or other study documentation.

Randomization will be carried out using real-time automated statistical software: eligible subjects will be randomly assigned to one of the two intervention arms (A, B) with a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Active smoker (≥ 30 packs/year)
* Former heavy smoker for ≤ 15 years (≥ 30 packs/year)
* Absence of tumors for at least 5 years
* Signature of informed consent for studio enrollment and processing of personal data

Exclusion Criteria:

* Severe chronic disease (e.g. severe respiratory and/or renal and/or hepatic and/or cardiac failure)
* Severe psychiatric problems
* Abuse of alcohol or other substances (including previous)

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7324 (Estimated)
Dates: Start 2022-09-17 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in lung cancer incidence | 3 years
  Change in lung cancer incidence: evaluate the impact on lung cancer incidence through LDCT at annual or biennial intervals.
Change in lung cancer specific and overall mortality | 5 years
  Change in lung cancer specific and overall mortality: evaluate the impact on lung cancer mortality through LDCT at annual or biennial intervals.
Change in smoking status | 3 years
  Change in the percentage of smokers
Molecular risk profile through assessing the value of microRNA in blood and tissue samples | 5 years
  MicroRNA expression profile, using TaqMan microfluidic cards: increased efficiency of lung cancer diagnosis by requiring less CT examinations while retaining the ability to diagnose lung cancer at curative state.

CONTACTS AND LOCATIONS:
Overall Officials: Ugo Pastorino, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Chiara Bovolenta, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pastorino U, Ladisa V, Trussardo S, Sabia F, Rolli L, Valsecchi C, Ledda RE, Milanese G, Suatoni P, Boeri M, Sozzi G, Marchiano A, Munarini E, Boffi R, Gallus S, Apolone G. Cytisine Therapy Improved Smoking Cessation in the Randomized Screening and Multiple Intervention on Lung Epidemics Lung Cancer Screening Trial. J Thorac Oncol. 2022 Nov;17(11):1276-1286. doi: 10.1016/j.jtho.2022.07.007. Epub 2022 Jul 28. PMID 35908731
- [Background] Milanese G, Sabia F, Ledda RE, Sestini S, Marchiano AV, Sverzellati N, Pastorino U. Volumetric Measurements in Lung Cancer Screening Reduces Unnecessary Low-Dose Computed Tomography Scans: Results from a Single-Center Prospective Trial on 4119 Subjects. Diagnostics (Basel). 2022 Jan 18;12(2):229. doi: 10.3390/diagnostics12020229. PMID 35204320
- [Background] Pastorino U, Boeri M, Sestini S, Sabia F, Milanese G, Silva M, Suatoni P, Verri C, Cantarutti A, Sverzellati N, Corrao G, Marchiano A, Sozzi G. Baseline computed tomography screening and blood microRNA predict lung cancer risk and define adequate intervals in the BioMILD trial. Ann Oncol. 2022 Apr;33(4):395-405. doi: 10.1016/j.annonc.2022.01.008. Epub 2022 Jan 25. PMID 35091076
- [Background] Silva M, Milanese G, Ledda RE, Nayak SM, Pastorino U, Sverzellati N. European lung cancer screening: valuable trial evidence for optimal practice implementation. Br J Radiol. 2022 May 1;95(1133):20200260. doi: 10.1259/bjr.20200260. Epub 2022 Jan 7. PMID 34995141
- [Background] Rundo L, Ledda RE, di Noia C, Sala E, Mauri G, Milanese G, Sverzellati N, Apolone G, Gilardi MC, Messa MC, Castiglioni I, Pastorino U. A Low-Dose CT-Based Radiomic Model to Improve Characterization and Screening Recall Intervals of Indeterminate Prevalent Pulmonary Nodules. Diagnostics (Basel). 2021 Sep 3;11(9):1610. doi: 10.3390/diagnostics11091610. PMID 34573951
- [Background] Tringali G, Milanese G, Ledda RE, Pastorino U, Sverzellati N, Silva M. Lung Cancer Screening: Evidence, Risks, and Opportunities for Implementation. Rofo. 2021 Oct;193(10):1153-1161. doi: 10.1055/a-1382-8648. Epub 2021 Mar 26. PMID 33772489
- [Background] Silva M, Milanese G, Sestini S, Sabia F, Jacobs C, van Ginneken B, Prokop M, Schaefer-Prokop CM, Marchiano A, Sverzellati N, Pastorino U. Lung cancer screening by nodule volume in Lung-RADS v1.1: negative baseline CT yields potential for increased screening interval. Eur Radiol. 2021 Apr;31(4):1956-1968. doi: 10.1007/s00330-020-07275-w. Epub 2020 Sep 30. PMID 32997182
- [Background] Pastorino U, Sverzellati N, Sestini S, Silva M, Sabia F, Boeri M, Cantarutti A, Sozzi G, Corrao G, Marchiano A. Ten-year results of the Multicentric Italian Lung Detection trial demonstrate the safety and efficacy of biennial lung cancer screening. Eur J Cancer. 2019 Sep;118:142-148. doi: 10.1016/j.ejca.2019.06.009. Epub 2019 Jul 20. PMID 31336289
- [Background] Pastorino U, Silva M, Sestini S, Sabia F, Boeri M, Cantarutti A, Sverzellati N, Sozzi G, Corrao G, Marchiano A. Prolonged lung cancer screening reduced 10-year mortality in the MILD trial: new confirmation of lung cancer screening efficacy. Ann Oncol. 2019 Oct 1;30(10):1672. doi: 10.1093/annonc/mdz169. No abstract available. PMID 31168572
- [Background] Pastorino U, Silva M, Sestini S, Sabia F, Boeri M, Cantarutti A, Sverzellati N, Sozzi G, Corrao G, Marchiano A. Prolonged lung cancer screening reduced 10-year mortality in the MILD trial: new confirmation of lung cancer screening efficacy. Ann Oncol. 2019 Jul 1;30(7):1162-1169. doi: 10.1093/annonc/mdz117. PMID 30937431
- [Background] Gallus S, Lugo A, Suatoni P, Taverna F, Bertocchi E, Boffi R, Marchiano A, Morelli D, Pastorino U. Effect of Tobacco Smoking Cessation on C-Reactive Protein Levels in A Cohort of Low-Dose Computed Tomography Screening Participants. Sci Rep. 2018 Aug 27;8(1):12908. doi: 10.1038/s41598-018-29867-9. PMID 30150729
- [Background] Silva M, Prokop M, Jacobs C, Capretti G, Sverzellati N, Ciompi F, van Ginneken B, Schaefer-Prokop CM, Galeone C, Marchiano A, Pastorino U. Long-Term Active Surveillance of Screening Detected Subsolid Nodules is a Safe Strategy to Reduce Overtreatment. J Thorac Oncol. 2018 Oct;13(10):1454-1463. doi: 10.1016/j.jtho.2018.06.013. Epub 2018 Jul 16. PMID 30026071
- [Background] Sozzi G, Boeri M, Rossi M, Verri C, Suatoni P, Bravi F, Roz L, Conte D, Grassi M, Sverzellati N, Marchiano A, Negri E, La Vecchia C, Pastorino U. Clinical utility of a plasma-based miRNA signature classifier within computed tomography lung cancer screening: a correlative MILD trial study. J Clin Oncol. 2014 Mar 10;32(8):768-73. doi: 10.1200/JCO.2013.50.4357. Epub 2014 Jan 13. PMID 24419137
- [Background] Pastorino U, Rossi M, Rosato V, Marchiano A, Sverzellati N, Morosi C, Fabbri A, Galeone C, Negri E, Sozzi G, Pelosi G, La Vecchia C. Annual or biennial CT screening versus observation in heavy smokers: 5-year results of the MILD trial. Eur J Cancer Prev. 2012 May;21(3):308-15. doi: 10.1097/CEJ.0b013e328351e1b6. PMID 22465911
- [Background] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641
- [Background] de Koning HJ, van der Aalst CM, de Jong PA, Scholten ET, Nackaerts K, Heuvelmans MA, Lammers JJ, Weenink C, Yousaf-Khan U, Horeweg N, van 't Westeinde S, Prokop M, Mali WP, Mohamed Hoesein FAA, van Ooijen PMA, Aerts JGJV, den Bakker MA, Thunnissen E, Verschakelen J, Vliegenthart R, Walter JE, Ten Haaf K, Groen HJM, Oudkerk M. Reduced Lung-Cancer Mortality with Volume CT Screening in a Randomized Trial. N Engl J Med. 2020 Feb 6;382(6):503-513. doi: 10.1056/NEJMoa1911793. Epub 2020 Jan 29. PMID 31995683
- [Background] Becker N, Motsch E, Trotter A, Heussel CP, Dienemann H, Schnabel PA, Kauczor HU, Maldonado SG, Miller AB, Kaaks R, Delorme S. Lung cancer mortality reduction by LDCT screening-Results from the randomized German LUSI trial. Int J Cancer. 2020 Mar 15;146(6):1503-1513. doi: 10.1002/ijc.32486. Epub 2019 Jun 20. PMID 31162856
- [Background] Quaife SL, Ruparel M, Dickson JL, Beeken RJ, McEwen A, Baldwin DR, Bhowmik A, Navani N, Sennett K, Duffy SW, Wardle J, Waller J, Janes SM. Lung Screen Uptake Trial (LSUT): Randomized Controlled Clinical Trial Testing Targeted Invitation Materials. Am J Respir Crit Care Med. 2020 Apr 15;201(8):965-975. doi: 10.1164/rccm.201905-0946OC. PMID 31825647
- See also: 4-IN THE LUNG RUN: towards INdividually tailored INvitations, screening INtervals, and INtegrated co-morbidity reducing strategies in lung cancer screening — https://cordis.europa.eu/project/id/848294
- See also: Cancer Intervention and Surveillance Modeling Network (CISNET) Lung Cancer Working Group. — https://www.ncbi.nlm.nih.gov/books/NBK568586/pdf/Bookshelf_NBK568586.pdf